CLINICAL TRIAL: NCT05050656
Title: "Preoperative Oral Duloxetine: Does it Affect Duration of Spinal Anesthesia and Early Postoperative Pain After Arthroscopic ACL Repair?" a Prospective, Randomized, Double-blind Controlled Trial
Brief Title: Oral Duloxetine as a Premedication for Postoperative Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Samir Abdelsalam, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FMASU R 63/ 2021
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (duloxetine group) (Active Comparator): Two hours before surgery, participants received oral duloxetine 60 mg tablets in the ward then transferred to OR to receive spinal anesthesia before surgery.
  Interventions: Drug: Duloxetine 60mg
- Group C (control group) (Placebo Comparator): Two hours before surgery, participants received oral placebo tablets in the ward then transferred to OR to receive spinal anesthesia before surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine 60mg — Duloxetine is a selective SNRI prescribed in depression, anxiety, and chronic pain like diabetic neuropathy and fibromyalgia, it acts through central and peripheral pain modulation
  Arms: Group D (duloxetine group)
Drug: Placebo — placebo tablets identical to duloxetine tablets
  Arms: Group C (control group)

SUMMARY:
The purpose of the study is to use duloxetine as premedication in Anterior cruciate ligament repair under spinal anesthesia and evaluate the effect on onset and duration of spinal anesthesia and postoperative pain control.

DETAILED DESCRIPTION:
We designed this randomized, double-blind study to evaluate the effectiveness of administration of oral duloxetine 2 hours preoperatively on the onset and the duration of the spinal anesthesia in arthroscopic anterior cruciate ligament (ACL) repair and the role of duloxetine on postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I or II.
* Sex: Both sexes.
* Age between 18 and 50.
* Height 155-180 cm.
* Patients scheduled for arthroscopic anterior cruciate ligament (ACL) repair under spinal anesthesia.

Exclusion Criteria:

* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* Had a history of drug or alcohol abuse.
* Taking opioids or sedative medications.
* Inability to communicate with patients to evaluate the postoperative pain.
* Need for postoperative ICU hospitalization.
* Hepatic or renal failure.
* Patients with a history of taking duloxetine or any SSRIs.
* Contraindications to regional anesthesia (including coagulopathy and local infection).
* Psychiatric disorders with antipsycotics or antidepressants (tricylic or MAOIs).
* Antiplatelets (aspirin, clopidogrel) or anticoagulant (warfarin).
* Quinolones (ciprofloxacin).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Assess the onset of spinal anesthesia | 20 min
  Time to T10 sensory block and time to Bromage 1 motor block

SECONDARY OUTCOMES:
Duration of spinal anesthesia | 4 hours
  Two-dermatomes regression for sensory recovery and return to Bromage 2 for motor recovery
Postoperative pain | 24 hours
  Will be assessed by the patient using the visual analog scale (VAS, 0=no pain; 10=worst possible pain) every 4hrs up to 24hrs after the operation.
Time for first postoperative rescue analgesia request, frequency, and total morphine consumption | 24 hours
  All participants will receive intravenous paracetamol, one gram every 8hrs, VAS score of 4 or more will receive 3 mg morphine intravenously and not be repeated more frequently than 4hrs limited to 12 mg morphine per 24hrs after operation

CONTACTS AND LOCATIONS:
Overall Officials: tamer abdelaziz, MD, Principal Investigator — Faculty of medicine, Ain Shams University, Cairo, Egypt
Locations (1):
- faculty of medicine, Ain Shams University, Cairo, Egypt